CLINICAL TRIAL: NCT06340841
Title: Lived Experiences Measured Using Ring Study: Single Session Intervention to Motivate Behavioral Change
Brief Title: LEMURS SSI: Evaluation of Behavioral Incentives
Acronym: LEMURSSI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Matthew Price, Professor, University of Vermont
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: LEMURS SSI 24
Record Dates: First submitted 2024-03-22; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Incentives

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four incentive conditions and receive rewards based on their completion of such activities. There are two main factors (Recipient x Restoration) that will create four distinct groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individual Receives Incentive - No Restorative Incentive (Experimental): Participant receives incentives directly
  Interventions: Behavioral: Personal Incentives
- Individual Receives Incentive -Restorative Incentive (Experimental): The participant receives incentives directly. There is a restorative incentive if they miss an activity.
  Interventions: Behavioral: Personal Restorative Incentives
- Charity Receives Incentive - No Restorative Incentive (Experimental): Participant earns money for charity
  Interventions: Behavioral: Charity Incentives
- Charity Receives Incentive -Restorative Incentive (Experimental): Participant earns money for charity. There is a restorative incentive if they miss an activity.
  Interventions: Behavioral: Charity Restorative Incentives

INTERVENTIONS:
Behavioral: Personal Incentives — The participant receives incentives directly if they complete an activity on a given day.
  Arms: Individual Receives Incentive - No Restorative Incentive
Behavioral: Personal Restorative Incentives — The participant receives incentives directly if they complete an activity on a given day. They are given an additional incentive to return to completing activities if they did not complete an activity on a prior day.
  Arms: Individual Receives Incentive -Restorative Incentive
Behavioral: Charity Incentives — The participant earns compensation for charity if they complete an activity on a given day.
  Arms: Charity Receives Incentive - No Restorative Incentive
Behavioral: Charity Restorative Incentives — The participant earns compensation for charity if they complete an activity on a given day. They are given an additional incentive for charity to return to completing activities if they did not complete an activity on a prior day.
  Arms: Charity Receives Incentive -Restorative Incentive

SUMMARY:
The goal of this substudy is to determine if a brief single-session-intervention (SSI) coupled with different incentive strategies to support engaging in wellness-related activities.

DETAILED DESCRIPTION:
The goal of this substudy is to determine if a brief single-session-intervention (SSI) coupled with different incentive strategies to support engaging in wellness-related activities. Participants will be given a brief SSI that will provide education and strategies to improve a wellness related goal (e.g., improve sleep, improve physical activity, improve mental health). They will then be asked to select a series of wellness related-behaviors in support of that goal to complete each day (e.g., going for a 20 minute walk, going to bed at a specific time). Participants will be randomized to one of four incentive conditions and receive rewards based on their completion of such activities. The aim of the study is to determine which incentive strategy may prove most effective in promoting wellness behaviors. There are two main factors (Recipient x Restoration) that will create four distinct groups. Recipient refers to who will receive the incentive - either an individual or a charity. Restoration refers to what happens when a participant misses a day of completing their goal - they are given a restorative (additional) incentive to participants on the following day or not given such an incentive. The primary hypothesis is that individuals receiving the incentive with a restorative element will result in significantly more activities completed. Additional hypotheses regarding differences among the other groups are not made given the lack of prior work on these strategies in this area.

ELIGIBILITY:
Inclusion Criteria:

Current undergraduate student in their first year of school own a mobile device

Exclusion Criteria:

None

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Activity Completion | up to 6 months
  Number of wellness activities completed

SECONDARY OUTCOMES:
Depression, Anxiety, Stress Scale - 21 | up to 6 months
  Summary Score on Depression Scale, higher scores indicate greater depression
Depression, Anxiety, Stress Scale - 21 | up to 6 months
  Summary Score on Anxiety Scale, higher scores indicate greater anxiety
Depression, Anxiety, Stress Scale - 21 | up to 6 months
  Summary Score on Stress Scale, higher scores indicate greater stress
Warwick-Edinburgh Mental Well-being Scale | up to 6 months
  Summary Score on the Measure, higher scores indicate better well-being
Oura Ring Sleep Index | up to 6 months
  Biometric Sleep recorded from an Oura Ring, higher scores indicate better sleep

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No